CLINICAL TRIAL: NCT00419913
Title: A Randomized Placebo-Controlled Trial of Dehydroepiandrosterone (DHEA) Treatment for Two Months Before Starting Ovulation Induction for in Vitro Fertilization (IVF)
Brief Title: A Trial of Dehydroepiandrosterone (DHEA) Treatment for in Vitro Fertilization (IVF)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Failure to recruit sufficient participants.
Sponsor: Center for Human Reproduction (Other)
Collaborators: Foundation for Reproductive Medicine (Other)
Responsible Party: Dr. David H. Barad, Center for Human Reproduction
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHR2006 1.0
Record Dates: First submitted 2007-01-07; First posted 2007-01-09 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Infertility; Decreased Ovarian Reserve
Keywords: Ovulation Induction; In vitro Fertilization; Pregnancy
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): Dehydroepiandrosterone (DHEA) 25mg tid
  Interventions: Dietary Supplement: Dehydroepiandrosterone
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Dehydroepiandrosterone

INTERVENTIONS:
Dietary Supplement: Dehydroepiandrosterone — DHEA 25 mg tid

SUMMARY:
Our long term goal is to elucidate the role of DHEA on follicular dynamics in the human ovary and to better understand the interaction of DHEA supplementation with other treatments for ovulation induction, especially among older reproductive age women.

The specific hypothesis behind the proposed research is that DHEA is a regulator of follicular dynamics acting in the early pre-gonadotropin dependent stage of initial primordial follicle recruitment and growth.

DETAILED DESCRIPTION:
Specific Aims:

The ability of women to respond to ovulation inducing medications also called ovarian reserve, declines with age. (Navot, Bergh et al. 1991; Scott, Leonardi et al. 1993; Toner and Flood 1993 ; Scott and Hofmann 1995; Scott 1996; ASRM 2002) When attempting in-vitro fertilization (IVF), older women produce few oocytes (Chuang, Chen et al. 2003; Orvieto, Bar-Hava et al. 2004) and yield few normal embryos, even when exposed to maximal gonadotropin stimulation.(Orvieto, Bar-Hava et al. 2004) As a result reproductive success for women over 40 years old is significantly reduced compared to younger women. Older ovaries have few antral follicles, high rates of follicular degeneration (atresia)(Faddy 2000) and increased "resistance" to ovulation induction.(Filicori 1999; Chuang, Chen et al. 2003; Kupesic, Kurjak et al. 2003) A delay in onset of atresia could salvage follicles for later ovulation.

Our long term goal is to elucidate the role of DHEA on follicular dynamics in the human ovary and to better understand the interaction of DHEA supplementation with other treatments for ovulation induction, especially among older reproductive age women.

The specific hypothesis behind the proposed research is that DHEA is a regulator of follicular dynamics acting in the early pre-gonadotropin dependent stage of initial primordial follicle recruitment and growth. That hypothesis is based on the following observations. First, at physiological doses DHEA increases serum levels of the insulin-like growth factor (IGF-l).(Casson, Santoro et al. 1998) DHEA is produced by the ovarian theca,(Burger 2002) increased concentration of follicular DHEA is associated with increased aromatase activity,(Franks, Mason et al. 2000) and DHEA is a prohormone that is converted in peripheral tissues to estrogens.(Haning, Hackett et al. 1993) Second, DHEA exposed rats simulate polycystic ovary syndrome (PCO)(Roy, Mahesh et al. 1962) and have a higher percentage of meiotically active oocytes and less evidence of atresia.(Anderson, Lee et al. 1997) Women chronically exposed to androgens can develop PCO-like ovaries.(Amirikia, Savoy-Moore et al. 1986) Women with anovulatory PCO have less evidence of follicle atresia.(Franks, Mason et al. 2000) Third, Casson et al (Casson, Lindsay et al. 2000) found a small increase in follicle number and E2 response to ovulation induction after two months of DHEA (80 mg/day) administration to five women, with proven ovarian resistance to stimulation.

Preliminary data Barad and Gleicher reported a patient with a history of severely decreased ovarian reserve who dramatically increased her oocyte production over nine cycles of treatment while taking DHEA and ovulation induction.(Barad and Gleicher 2005) The dramatic increase in oocyte production seen in this patient did not occur until after four months of DHEA treatment (75 mg/day). This treatment duration is in keeping with the interval required for normal follicular initiation of recruitment and growth(Gougeon 1986) and raises that possibility that the Casson et al. did not treat their subjects long enough to achieve maximum effect. Our case report was followed by a case control study that showed increased oocyte production and improved embryo quality among 25 DHEA treated patients, whose pre-treatment cycle acted as control.(Barad and Gleicher 2005)

More recently we showed that DHEA treated patients with significant decreased ovarian reserve have higher pregnancy rates compared to controls.(Barad, Brill et al. 2006)

Based on these observations the experimental focus of this project is on the interaction of DHEA adjuvant treatment with gonadotropin treatment during ovulation induction. The specific aims are designed to provide a comprehensive assessment of this effect.

1. DHEA treatment will increase pregnancy rates among women 40 to 45 years old.
2. DHEA treatment will increase antral follicle counts.
3. DHEA will lead to increased anti-mullerian (AMH) hormone levels.
4. DHEA treatment will increase mean and peak follicular phase estradiol.
5. DHEA treatment will increase the number of oocytes retrieved in IVF cycles compared to placebo.

Research Plan:

Placebo controlled randomized trial of 2 months of DHEA pretreatment prior to ovulation induction for IVF-ET.

Hypothesis 1:

Two months of DHEA pretreatment will improve the chance of pregnancy and lead to greater oocyte and embryo yields relative to placebo treated control patients.

Hypothesis 2:

Embryos produced following 2 months of pretreatment with either DHEA alone OR with DHEA plus supplemental FSH 150 units per day will result in embryos with better morphology

Hypothesis 3a-c:

Two months of DHEA pretreatment will result in: a) increased antral follicle counts, increased AMH, b) increased mean and peak estradiol and c) increased oocyte production

Recruitment plan:

* New patients presenting for treatment.
* Possible print, magazine or Radio advertisement

References:

Amirikia, H., R. T. Savoy-Moore, et al. (1986). "The effects of long-term androgen treatment on the ovary." Fertil Steril 45(2): 202-8.

Anderson, E., G. Y. Lee, et al. (1997). "Polycystic ovarian condition in the dehydroepiandrosterone-treated rat model: hyperandrogenism and the resumption of meiosis are major initial events associated with cystogenesis of antral follicles." Anat Rec 249(1): 44-53.

ASRM (2002). "Aging and infertility in women: a committee opinion." Fertil Steril 78(1): 215-9.

Barad, D., H. Brill, et al. (2006). "Dehydroepiandrosterone (DHEA) Increases Pregnancy Rates in Women with Diminished Ovarian Reserve:

A Case Controlled Study." Submitted for Publication. Barad, D. and N. Gleicher (2005). "Effect of dehydroepiandrosterone (DHEA) on oocyte and embryo yields, embryo grade and cell number in IVF." Human Reproduction In Press.

Barad, D. and N. Gleicher (2005). "Increased Oocyte Production after Treatment with Dehydroepiandrosterone." Fertil Steril 84(3): 756.

Burger, H. G. (2002). "Androgen production in women." Fertil Steril 77 Suppl 4: S3-5.

Casson, P. R., M. S. Lindsay, et al. (2000). "Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series." Hum Reprod 15(10): 2129-32.

Casson, P. R., N. Santoro, et al. (1998). "Postmenopausal dehydroepiandrosterone administration increases free insulin-like growth factor-I and decreases high-density lipoprotein: a six-month trial." Fertil Steril 70(1): 107-10.

Chuang, C. C., C. D. Chen, et al. (2003). "Age is a better predictor of pregnancy potential than basal follicle-stimulating hormone levels in women undergoing in vitro fertilization." Fertil Steril 79(1): 63-8.

Faddy, M. J. (2000). "Follicle dynamics during ovarian ageing." Mol Cell Endocrinol 163(1-2): 43-8.

Filicori, M. (1999). "The role of luteinizing hormone in folliculogenesis and ovulation induction." Fertil Steril 71(3): 405-14.

Franks, S., H. Mason, et al. (2000). "Follicular dynamics in the polycystic ovary syndrome." Mol Cell Endocrinol 163(1-2): 49-52.

Gougeon, A. (1986). "Dynamics of follicular growth in the human: a model from preliminary results." Hum Reprod 1(2): 81-7.

Haning, R. V., Jr., R. J. Hackett, et al. (1993). "Plasma dehydroepiandrosterone sulfate serves as a prehormone for 48% of follicular fluid testosterone during treatment with menotropins." J Clin Endocrinol Metab 76(5): 1301-7.

Kupesic, S., A. Kurjak, et al. (2003). "Three-dimensional ultrasonographic ovarian measurements and in vitro fertilization outcome are related to age." Fertil Steril 79(1): 190-7.

Navot, D., P. A. Bergh, et al. (1991). "Poor oocyte quality rather than implantation failure as a cause of age-related decline in female fertility." Lancet 337(8754): 1375-7.

Orvieto, R., I. Bar-Hava, et al. (2004). "Results of in vitro fertilization cycles in women aged 43-45 years." Gynecol Endocrinol 18(2): 75-8.

Roy, S., V. Mahesh, et al. (1962). "The effect of dehydroepiandrosterone and D4-androstenedione on the reproductive organs of female rats: Production of cystic changes in the ovary." Nature 196: 42-43.

Scott, R. T., Jr. (1996). "Evaluation and treatment of low responders." Semin Reprod Endocrinol 14(4): 317-37.

Scott, R. T., Jr. and G. E. Hofmann (1995). "Prognostic assessment of ovarian reserve." Fertil Steril 63(1): 1-11.

Scott, R. T., M. R. Leonardi, et al. (1993). "A prospective evaluation of clomiphene citrate challenge test screening of the general infertility population." Obstet Gynecol 82(4 Pt 1): 539-44.

Toner, J. P. and J. T. Flood (1993). "Fertility after the age of 40." Obstet Gynecol Clin North Am 20(2): 261-72.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 40 and less than 45 years old presenting for IVF treatment.
* Willingness to sign informed consent for study randomization.
* Willingness to participate in 2 months pre-IVF treatment.

Exclusion Criteria:

* Medical condition that would contraindicate pregnancy, ovulation induction or general anesthesia.
* Family history of significant genetic disease, or factor V Leiden thrombophilia.
* Inability to present for monitoring visits.
* Inability to follow medication instruction.

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy per cycle of treatment | 1 year

SECONDARY OUTCOMES:
Embryos per cycle of treatment | 1 year
Oocytes per cycle of treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Barad, MD, Principal Investigator — Center for Human Reproduction
Locations (2):
- Center for Human Reproduction, New York, New York, United States
- Institute fur Reproduktionsmedzin und Endokrinologie, Bregenz, Austria

REFERENCES:
- [Background] Barad D, Gleicher N. Effect of dehydroepiandrosterone on oocyte and embryo yields, embryo grade and cell number in IVF. Hum Reprod. 2006 Nov;21(11):2845-9. doi: 10.1093/humrep/del254. Epub 2006 Sep 22. PMID 16997936
- [Background] Barad DH, Gleicher N. Increased oocyte production after treatment with dehydroepiandrosterone. Fertil Steril. 2005 Sep;84(3):756. doi: 10.1016/j.fertnstert.2005.02.049. PMID 16169414